CLINICAL TRIAL: NCT07321002
Title: Assessment of a Novel Shape-Adaptive Catheter With for Both Single-Shot and Large-Focal Pulsed Field Ablation the DePolar Mapping System in Persistent Atrial Fibrillation
Brief Title: PFLotus With the DePolar Mapping System in Patients With Persistent Atrial Fibrillation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Hanxiong Liu, Professor, The Third People's Hospital of Chengdu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFLotus with DePolar
Record Dates: First submitted 2025-12-09; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation; pulse field ablation; pulmonary vein isolaiton; left atrial posterior wall; mitral isthmus isolaiton; cavotricuspid isthmus isolation; superior vena cava; coronary sinus; epicardial ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation Group (Experimental): PVI and additional ablation strategies-including ablation of the left atrial posterior wall (LAPW), mitral isthmus (MI), cavotricuspid isthmus (CTI), and superior vena cava (SVC)-were performed in all patients with PerAF.
  Interventions: Device: Ablation with the PFLotus catheter and Depolar system

INTERVENTIONS:
Device: Ablation with the PFLotus catheter and Depolar system — PVI and additional ablation strategies-including ablation of the left atrial posterior wall (LAPW), mitral isthmus (MI), cavotricuspid isthmus (CTI), and superior vena cava (SVC)-were performed in all patients with PerAF using the PFLotus PFA catheter and Depolar mapping system.

SUMMARY:
This clinical trial aims to evaluate the safety and efficacy of pulmonary vein isolation (PVI), focal, and linear ablation in patients with persistent atrial fibrillation (PersAF) using a novel shape-adaptive pulsed field ablation (PFA) catheter (PFLotus, EnChannel Medical) integrated with a novel mapping system (DePolar, EnChannel Medical).

The primary study objectives are to determine:

* The incidence of serious procedure- or device-related adverse events within 7 days post-procedure (primary safety endpoint).
* The clinical effectiveness of the integrated PFA and mapping system.
* The ability of the novel PFA system to produce durable ablation lesions.

PersAF patients will be treated under general anesthesia using the PFLotus PFA catheter (bipolar, biphasic waveform; 850 V, 60 μs per pulse). Ablation targets, including PVI and other lesions (left atrial posterior wall, mitral isthmus, cavotricuspid isthmus, and superior vena cava), will be accessed under fluoroscopic and DePolar mapping system guidance.

Participants will:

1. Receive PVI, focal, and linear ablation using the PFLotus PFA catheter and DePolar mapping system under general anesthesia;
2. Be monitored for serious procedure- or device-related adverse events during the first 7 days post-procedure;
3. Undergo repeat electrophysiological mapping at 3 months to assess lesion durability;
4. Attend scheduled follow-up visits at 7 days, 30 days, and 3, 6, and 12 months post-ablation. Atrial arrhythmia recurrence will be assessed via 12-lead electrocardiography at each visit and by 24-hour or 7-day Holter monitoring at the 6- and 12-month visits.

DETAILED DESCRIPTION:
Background Atrial fibrillation (AF) is the most common persistent cardiac arrhythmia worldwide, affecting an estimated 1.5-2.0% of the general population. As the population ages, the prevalence of AF continues to rise, imposing a substantial and growing burden on healthcare systems. AF significantly impairs quality of life, elevates stroke risk fivefold, triples the incidence of heart failure, and increases overall mortality.

Initial AF management typically involves pharmacotherapy for rate control or rhythm control. Compared to antiarrhythmic drugs (AADs), catheter ablation offers superior efficacy in reducing AF recurrence, lowering cardiovascular hospitalization rates, and preventing arrhythmia relapse. The cornerstone of catheter ablation is pulmonary vein isolation (PVI), which electrically isolates the pulmonary veins from the left atrium. Current guidelines recommend catheter ablation, primarily PVI, for patients with symptomatic, drug-refractory paroxysmal AF, establishing it as a standard therapy for symptomatic paroxysmal or persistent AF.

Pulsed field ablation (PFA) induces cardiomyocyte death via irreversible electroporation using high-voltage, ultra-rapid electric fields. As a non-thermal energy modality, PFA demonstrates selective myocardial tissue affinity. This characteristic may enable durable lesion formation while sparing adjacent critical structures such as the esophagus, blood vessels, pulmonary veins, and phrenic nerve. Notably, PFA has not been associated with thermal energy complications like atrio-esophageal fistula, phrenic nerve palsy, or pulmonary vein stenosis, suggesting the potential for enhanced efficacy with an improved safety profile.

Recent evidence indicates that integrating three-dimensional (3D) mapping and navigation systems into PFA procedures can reduce radiation exposure while improving procedural accuracy and clinical outcomes.

Therefore, this study aims to evaluate the safety and efficacy of PVI, focal, and linear ablation in patients with persistent AF (PersAF) using a novel shape-adaptive PFA catheter (PFLotus, EnChannel Medical) integrated with a new mapping system (DePolar, EnChannel Medical).

Methods Study Population Eligible patients were aged 18-75 years with documented symptomatic persistent AF (duration 7-365 days) who were refractory or intolerant to at least one Class I or III antiarrhythmic drug.

Procedural Workflow All procedures were performed under general anesthesia. Activated clotting time was maintained at ≥300 seconds. An electroanatomic map of the left atrium and pulmonary veins was created using the PFLotus catheter and the DePolar system.

PVI and additional ablation strategies-including ablation of the left atrial posterior wall (LAPW), mitral isthmus (MI), cavotricuspid isthmus (CTI), and superior vena cava (SVC)-were performed in all patients. For MI ablation, if persistent epicardial connections were identified, adjunctive ablation within the coronary sinus was performed. After a 20-minute waiting period, isolation and block were reassessed.

Follow-up Post-ablation antiarrhythmic drug use was determined by the operator and typically discontinued after three months. Oral anticoagulation was maintained per guidelines. Structured follow-up was conducted at 7 days and 3 months post-ablation, with lesion durability assessed via invasive remapping at 3 months. Additional visits were scheduled at 6 and 12 months. Atrial tachyarrhythmia recurrence was assessed using 12-lead ECGs at each visit and 24-hour or 7-day Holter monitoring at 3, 6, and 12 months.

Endpoints The primary safety endpoint was the incidence of primary adverse events (PAEs) within 7 days post-ablation. Later-occurring events-including device- or procedure-related death, atrio-esophageal fistula, and PV stenosis-were also classified as PAEs. Persistent diaphragmatic paralysis or phrenic nerve palsy at 3 months was considered a PAE.

The primary efficacy endpoint was acute procedural success, defined as the proportion of patients achieving: 1) complete electrical isolation of all pulmonary veins, and 2) confirmed bidirectional block at all targeted linear ablation sites (LAPW, MI, CTI, and SVC) in patients undergoing such ablation.

Secondary efficacy endpoints included:

1. Acute PV isolation success rate.
2. Acute success rate of bidirectional block for each linear ablation site.
3. Durable success rate of bidirectional block for each linear ablation site at 3-month remapping.
4. One-year freedom from atrial tachyarrhythmia recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years (inclusive). 2. Diagnosis of symptomatic persistent atrial fibrillation (AF), defined as documented AF episodes exceeding 7 days or a documented history of persistent AF. Additionally, at least one of the following criteria must be met within 365 days prior to enrollment:

1. A 24-hour ambulatory ECG (Holter) recording demonstrating AF throughout the entire monitoring period.
2. Two separate standard 12-lead ECGs, taken at least 7 days apart, both confirming AF.

3. Documented failure or intolerance to at least one Class I or Class III antiarrhythmic drug (AAD).

4. Willingness to participate in the trial, ability to comply with protocol-specified follow-up assessments, and provision of written informed consent.

Exclusion Criteria:

1. Paroxysmal atrial fibrillation (AF)；
2. AF caused by electrolyte disorders, thyroid diseases, or reversible/non-cardiac etiologies；
3. Patients undergoing retreatment after ablation for rapid atrial tachyarrhythmias；
4. Patients with sustained ventricular tachycardia or ventricular fibrillation；
5. Left atrial anteroposterior diameter > 55 mm；
6. Pulmonary vein (PV) stenosis (>70%) or prior PV stent implantation；
7. History of left atrial ablation or cardiac surgery (including left atrial appendage closure)；
8. Implantation of permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardioverter-defibrillator (with or without biventricular pacing function)；
9. Contraindications to anticoagulation, or history of coagulation or bleeding abnormalities；
10. Severe pulmonary disease: severe pulmonary arterial hypertension or any pulmonary disease with severe dyspnea involving blood gas abnormalities；
11. Any of the following cardiac surgeries, implants, or conditions:

    * Prosthetic heart valve
    * NYHA Class III or IV congestive heart failure, or left ventricular ejection fraction (LVEF) < 40%
    * Atrial septal defect or ventricular septal defect closure
    * Atrial myxoma, left atrial appendage device implantation or occlusion
12. History of any of the following within 3 months prior to the procedure:

    * Myocardial infarction
    * Unstable angina
    * Percutaneous coronary intervention
    * Cardiac surgery (including coronary artery bypass grafting)
    * Hospitalization for heart failure
    * Pericarditis
13. History of any of the following within 3 months prior to the procedure:

    * Cerebral infarction or transient ischemic attack (TIA)
    * Documented thromboembolic events (e.g., confirmed by transesophageal echocardiography [TEE])
14. History of malignant tumor or expected life expectancy < 12 months；
15. Mental disorders or history of mental illness with inability to cooperate independently；
16. Lactating, pregnant, or women planning or potentially becoming pregnant；
17. Acute or severe systemic infection, or significant abnormalities in liver/renal function；
18. Participation in other interventional clinical trials, or ineligibility for enrollment as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Primary Adverse Events (PAEs) Within 3 Months Post-Ablation [Primary Safety Endpoint] | Within 3 months post the index ablation
  The primary safety endpoint is defined as the incidence of primary adverse events (PAEs) in patients within 3 months after the index ablation. PAEs include: ① Adverse events occurring within 7 days post-ablation; ② Later-occurring events (device- or procedure-related death, atrio-esophageal fistula, pulmonary vein [PV] stenosis);
  ③ Persistent diaphragmatic paralysis or phrenic nerve palsy at 3 months post-ablation.
Rate of Acute Procedural Success: Complete Pulmonary Vein Isolation and Bidirectional Block at Targeted Linear Ablation Sites [Primary Efficacy Endpoint] | Immediate after the ablation procedure
  The primary efficacy endpoint is defined as the rate of acute procedural success immediately after the ablation procedure. Acute procedural success is confirmed when patients meet the following criteria:
  1. Complete electrical isolation of all pulmonary veins;
  2. Bidirectional block verified at all targeted linear ablation sites (including left atrial posterior wall [LAPW], mitral isthmus [MI], cavotricuspid isthmus [CTI], and superior vena cava [SVC]) in those undergoing linear ablation.

SECONDARY OUTCOMES:
Rate of Acute Pulmonary Vein (PV) Isolation Success [Secondary Efficacy Endpoint] | Immediate after the index ablation procedure
  Defined as the proportion of participants who achieve complete electrical isolation of all targeted pulmonary veins immediately after the index ablation procedure.
Acute Bidirectional Block Success Rate for Each Targeted Linear Ablation Site [Secondary Efficacy Endpoint] | Immediate after the index ablation procedure
  Defined as the proportion of each targeted linear ablation site (LAPW, MI, CTI, SVC) that achieves verified bidirectional block immediately after the index ablation procedure. Each linear site is assessed independently, and the success rate for each site is reported separately.
Durable Bidirectional Block Success Rate for Each Targeted Linear Ablation Site at 3-Month Remapping [Secondary Efficacy Endpoint] | 3 months post the index ablation procedure
  Defined as the proportion of each targeted linear ablation site (LAPW, MI, CTI, SVC) that maintains verified bidirectional block (without recurrence of conduction) at 3-month remapping after the index ablation procedure. Each linear site is assessed independently, and the durable success rate for each site is reported separately.
1-Year Freedom from Atrial Tachyarrhythmia Recurrence [Secondary Efficacy Endpoint] | 1 year post the index ablation procedure
  Defined as the proportion of participants who remain free from recurrent atrial tachyarrhythmias (including atrial fibrillation, atrial flutter, atrial tachycardia) within 1 year after the index ablation procedure. Recurrence is defined as any episode of atrial tachyarrhythmia lasting ≥30 seconds, confirmed by 12-lead electrocardiogram or 72-hour Holter monitoring, after the 3-month blanking period.

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD to be shared include baseline demographic and clinical data, procedural parameters, safety data (adverse events within 7 days and follow-up), effectiveness data, and post-PFA voltage mapping results. These IPD are all data used in the primary results publication, as sharing them supports reproducible research and advances the understanding of PFLotus PFA Catheters and Depolar mapping system in persistent AF.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2-year post the primary publication
Access Criteria: 1. Eligible Recipients Qualified researchers with academic/institutional affiliation, who submit a feasible research proposal and agree to comply with data protection regulations.
  2. Accessible Materials De-identified individual participant data (baseline, procedural, follow-up data related to PFA/AF) and supporting documents (study protocol, statistical analysis plan, redacted clinical study report). Identifiable information and raw imaging data are excluded.
  3. Access Process Submit application (proposal, CV, IRB approval, signed DUA) to the corresponding author via designated email.